CLINICAL TRIAL: NCT01378273
Title: Preterm Erythropoietin Neuroprotection Trial (PENUT Trial)
Acronym: PENUT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Sandra Juul, Professor of Pediatrics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00007464; U01NS077953 (NIH)
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Extreme Prematurity
Keywords: neuroprotection; erythropoietin; Epo; ELGANs; preterm; neonate
MeSH Terms: conditions — Premature Birth | interventions — Eosinophil Peroxidase; Erythropoietin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Subjects will receive 6 doses of vehicle intravenously during the first 2 weeks of life. Doses will be administered at 48 hour intervals from the time of enrollment. Following high dose administration, sham subcutaneous injections will be given three times a week through to 32-6/7 weeks postmenstrual age.
  Interventions: Other: Control
- Epo 1000 U/kg followed by 400 U/kg (Experimental): Subjects will receive 6 doses of intravenous Epo 1000 U/kg/dose at 48 hour intervals from the time of enrollment. Following the high dose period, subjects will receive subcutaneous Epo 400 U/kg/dose three times a week until 32-6/7 weeks postmenstrual age.
  Interventions: Drug: Epo

INTERVENTIONS:
Drug: Epo — Enrollment will occur within 24 hours of birth. Study drug will be administered intravenously for the first 6 doses. Subjects in the Epo arm will then receive 400 U/kg/dose three times a week until they reach 32-6/7 weeks postmenstrual age. Control infants will receive sham injections.
  Other Names: Epotin; Erythropoietin
  Arms: Epo 1000 U/kg followed by 400 U/kg
Other: Control — Subjects will receive 6 doses of vehicle intravenously during the first 2 weeks of life. Doses will be administered at 48 hour intervals from the time of enrollment. Following high dose administration, sham subcutaneous injections will be given three times a week through to 32-6/7 weeks postmenstrual age.
  Other Names: Saline
  Arms: Control

SUMMARY:
Recombinant human erythropoietin (Epo) is a promising novel neuroprotective agent. Epo decreases neuronal programmed cell death resulting from brain injury; it has anti-inflammatory effects, increases neurogenesis, and protects oligodendrocytes from injury.

We hypothesize that neonatal Epo treatment of ELGANs will decrease the combined outcome of death or severe NDI from 40% to 30% (primary outcome), or the combined outcome of death plus moderate or severe NDI from 60% to 40% (secondary outcome) measured at 24-26 months corrected age.

1. To determine whether Epo decreases the combined outcome of death or NDI at 24-26 months corrected age. NDI is defined as the presence of any one of the following: CP, Bayley Scales of Infant and Toddler Development, 3rd Edition (Bayley-III) Cognitive Scale < 70 (severe, 2 SD below mean) or 85 (moderate, 1 SD below mean). CP will be diagnosed and classified by standardized neurologic exam, with severity classified by Gross Motor Function Classification System (GMFCS).
2. To determine whether there are risks to Epo administration in ELGANs by examining, in a blinded manner, Epo-related safety measures comparing infants receiving Epo with those given placebo.
3. To test whether Epo treatment decreases serial measures of circulating inflammatory mediators, and biomarkers of brain injury.
4. To compare brain structure (as measured by MRI) in Epo treatment and control groups at 36 weeks PMA. MRI assessments will include documentation of intraventricular hemorrhage (IVH), white matter injury (WMI) and hydrocephalus (HC), volume of total and deep gray matter, white matter and cerebellum, brain gyrification, and tract-based spatial statistics (TBSS based on diffusion tensor imaging). As an exploratory aim, we will determine which of the above MRI measurements best predict neurodevelopment (CP, cognitive and motor scales) at 24-26 months corrected age.

Anticipated outcomes: Early Epo treatment of ELGANs will decrease biochemical and MRI markers of brain injury, will be safe, and will confer improved neurodevelopmental outcome at 24-26 months corrected age compared to placebo, and will provide a much-needed therapy for this group of vulnerable infants.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, study of Epo treatment of preterm infants 24-0/7 to 27-6/7 weeks of gestation, beginning in the first 24 hours after birth. Randomization will be stratified by site and gestational age at birth (<26 week or 26-27-6/7). Study size sample is 940 patients. We expect to evaluate 752 subjects at 24-26 months corrected age, our primary endpoint. There is no enrollment restriction based on gender, ethnicity or race. Enrollment is expected to take 24-26 months, with each subject participating through 24-26 months corrected age when neurodevelopmental outcomes are assessed. The combined outcome of death or severe NDI will be compared between Epo-treated and control subjects. All outcomes will be collected in a blinded manner. Subjects will be randomized by the data-coordinating center (DCC) to Epo treatment or placebo, and Epo treatment will continue until 32-6/7 weeks post menstrual age. Serial measurements of circulating inflammatory mediators and biomarkers of brain injury will be made. A brain MRI will be done at 36 weeks post menstrual age in the same subset of infants. Phone contact will occur at 4, 8, 12, and 18 months. Face to face follow up will occur at 24-26 months corrected age. The primary outcome is death or severe NDI at 24-26 months corrected age, with a secondary outcome of death or moderate NDI. Our primary sample size calculation is based on the conservative assumptions that Epo treatment will result in a 40% reduction in the severe NDI rate (the range in animal studies is 49-70%) and minimal impact on death. This would yield a control group rate for the primary outcome of 40.4% and an expected treated rate of 31.5% thus yielding an 8.9% lower rate of Death + NDI.

Clinical information including co-morbidities of extreme prematurity, information about transfusions, and specific laboratory values were collected in the PENUT database.

ELIGIBILITY:
Inclusion Criteria:

1. NICU inpatients between 24-0/7 and 27-6/7 weeks of gestation
2. Less than twenty four hours of age
3. Parental informed consent

Exclusion Criteria:

1. Major life-threatening anomalies (brain, cardiac, chromosomal anomalies)
2. Hematologic crises such as DIC, or hemolysis due to blood group incompatibilities
3. Polycythemia (hematocrit > 65)
4. Congenital infection

Ages: 24 Weeks to 27 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 941 (Actual)
Dates: Start 2013-12; Primary Completion 2019-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra E Juul, MD, PhD, Principal Investigator — University of Washington
Locations (19):
- United States (19):
  - University of Arkansas, Little Rock, Arkansas
  - University of Florida, Gainesville, Florida
  - South Miami Hospital, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - All Childrens Hospital, St. Petersburg, Florida
  - Prentice Women's Hospital, Chicago, Illinois
  - Children's Hospital of the University of Illinois, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Hospital, Boston, Massachusetts
  - Children's Hospital of Minnesota, MN, Minneapolis, Minnesota
  - University of Minnesota Amplatz Children's Hospital, Minneapolis, Minnesota
  - Children's Hospital of Minnesota, St. Paul, Saint Paul, Minnesota
  - University of New Mexico Children's Hospital, Albuquerque, New Mexico
  - Maia Fareri Children's Hospital, Valhalla, New York
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Methodist Children's Hospital, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available through the NINDS Data Archive: https://www.ninds.nih.gov/Current-Research/Research-Funded-NINDS/Clinical-Research/Archived-Clinical-Research-Datasets. The data will be de-identified and a limited access data set will be available after December 2020 through a request form on that page. Data dictionaries, in addition to study protocol, the statistical analysis plan, and the informed consent form will be included. The data will be made available upon publication of all PENUT Trial related manuscripts to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: December 2020
Access Criteria: The data will be made available upon publication of all PENUT Trial related manuscripts to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal.
URL: https://www.ninds.nih.gov/Current-Research/Research-Funded-NINDS/Clinical-Research/Archived-Clinical-Research-Datasets

REFERENCES:
- [Result] Juul SE, Mayock DE, Comstock BA, Heagerty PJ. Neuroprotective potential of erythropoietin in neonates; design of a randomized trial. Matern Health Neonatol Perinatol. 2015 Dec 2;1:27. doi: 10.1186/s40748-015-0028-z. eCollection 2015. PMID 27057344
- [Result] Starr MC, Askenazi DJ, Goldstein SL, MacDonald JW, Bammler TK, Afsharinejad Z, D Brophy P, Juul SE, Mayock DE, Hingorani SR. Impact of processing methods on urinary biomarkers analysis in neonates. Pediatr Nephrol. 2018 Jan;33(1):181-186. doi: 10.1007/s00467-017-3779-0. Epub 2017 Aug 19. PMID 28821985
- [Result] Juul SE, Comstock BA, Wadhawan R, Mayock DE, Courtney SE, Robinson T, Ahmad KA, Bendel-Stenzel E, Baserga M, LaGamma EF, Downey LC, Rao R, Fahim N, Lampland A, Frantz ID III, Khan JY, Weiss M, Gilmore MM, Ohls RK, Srinivasan N, Perez JE, McKay V, Vu PT, Lowe J, Kuban K, O'Shea TM, Hartman AL, Heagerty PJ; PENUT Trial Consortium. A Randomized Trial of Erythropoietin for Neuroprotection in Preterm Infants. N Engl J Med. 2020 Jan 16;382(3):233-243. doi: 10.1056/NEJMoa1907423. PMID 31940698
- [Derived] Hanna M, Chock VY, Kamath N, Raj A, Swanson JR, Griffin R, Askenazi DJ, Nesargi S. Acute Kidney Injury and Neurodevelopmental Outcomes in Extremely Premature Neonates: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Nov 3;8(11):e2543270. doi: 10.1001/jamanetworkopen.2025.43270. PMID 41222934
- [Derived] Valentine GC, Brandon OC, Perez KM, Strobel KM, Mayock DE, Law JB, Neches S, German K, Kolnik S, Heagerty PJ, Wood TR, Juul SE. Time to regain birthweight and in-hospital outcomes among United States-born extremely preterm newborns. Pediatr Res. 2025 Nov 10. doi: 10.1038/s41390-025-04563-3. Online ahead of print. PMID 41214292
- [Derived] Valentine GC, Perez KM, Wood TR, Mayock DE, Law JB, Kolnik S, Strobel KM, Brandon OC, Comstock BA, Heagerty PJ, Juul SE. Time to regain birthweight and association with neurodevelopmental outcomes among extremely preterm newborns. J Perinatol. 2024 Apr;44(4):554-560. doi: 10.1038/s41372-024-01869-8. Epub 2024 Jan 9. PMID 38195922
- [Derived] Strobel KM, Wood TR, Valentine GC, German KR, Gogcu S, Hendrixson DT, Kolnik SE, Law JB, Mayock DE, Comstock BA, Heagerty PJ, Juul SE. Contemporary definitions of infant growth failure and neurodevelopmental and behavioral outcomes in extremely premature infants at two years of age. J Perinatol. 2024 Jun;44(6):811-818. doi: 10.1038/s41372-023-01852-9. Epub 2024 Jan 9. PMID 38195921
- [Derived] Hingorani SR, Schmicker RH, Halloran B, Brophy P, Heagerty PJ, Juul S, Goldstein SL, Askenazi D; PENUT Investigators. Association Between Urinary Biomarkers and CKD in Extremely Low Gestational Age Neonates. Am J Kidney Dis. 2024 Apr;83(4):497-507. doi: 10.1053/j.ajkd.2023.09.008. Epub 2023 Nov 4. PMID 37926336
- [Derived] Valentine G, Perez K, Wood T, Mayock D, Law J, Kolnik S, Strobel K, Brandon O, Comstock B, Heagerty P, Juul S. Time to Regain Birthweight and Association with Neurodevelopmental Outcomes among Extremely Preterm Newborns. Res Sq [Preprint]. 2023 Sep 14:rs.3.rs-3249598. doi: 10.21203/rs.3.rs-3249598/v1. PMID 37790304
- [Derived] Starr MC, Griffin RL, Harer MW, Soranno DE, Gist KM, Segar JL, Menon S, Gordon L, Askenazi DJ, Selewski DT. Acute Kidney Injury Defined by Fluid-Corrected Creatinine in Premature Neonates: A Secondary Analysis of the PENUT Randomized Clinical Trial. JAMA Netw Open. 2023 Aug 1;6(8):e2328182. doi: 10.1001/jamanetworkopen.2023.28182. PMID 37561461
- [Derived] Starr MC, Griffin R, Gist KM, Segar JL, Raina R, Guillet R, Nesargi S, Menon S, Anderson N, Askenazi DJ, Selewski DT; Neonatal Kidney Collaborative Research Committee. Association of Fluid Balance With Short- and Long-term Respiratory Outcomes in Extremely Premature Neonates: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2248826. doi: 10.1001/jamanetworkopen.2022.48826. PMID 36580332
- [Derived] Hingorani S, Schmicker R, Ahmad KA, Frantz ID, Mayock DE, La Gamma EF, Baserga M, Khan JY, Gilmore MM, Robinson T, Brophy P, Heagerty PJ, Juul SE, Goldstein S, Askenazi D; PENUT Trial Consortium; PENUT Primary Investigators and coauthors. Prevalence and Risk Factors for Kidney Disease and Elevated BP in 2-Year-Old Children Born Extremely Premature. Clin J Am Soc Nephrol. 2022 Aug;17(8):1129-1138. doi: 10.2215/CJN.15011121. Epub 2022 Jul 19. PMID 35853728
- [Derived] Garcia MR, Comstock BA, Patel RM, Tolia VN, Josephson CD, Georgieff MK, Rao R, Monsell SE, Juul SE, Ahmad KA; PENUT Trial Consortium. Iron supplementation and the risk of bronchopulmonary dysplasia in extremely low gestational age newborns. Pediatr Res. 2023 Feb;93(3):701-707. doi: 10.1038/s41390-022-02160-2. Epub 2022 Jun 20. PMID 35725917
- [Derived] Valentine GC, Perez KM, Wood TR, Mayock DE, Comstock BA, Puia-Dumitrescu M, Heagerty PJ, Juul SE. Postnatal maximal weight loss, fluid administration, and outcomes in extremely preterm newborns. J Perinatol. 2022 Aug;42(8):1008-1016. doi: 10.1038/s41372-022-01369-7. Epub 2022 Mar 25. PMID 35338252
- [Derived] Askenazi DJ, Halloran BA, Heagerty PJ, Schmicker RH, Brophy P, Juul SE, Hingorani S, Goldstein SL; PENUT Trial Consortium. Gestational age, sex, and time affect urine biomarker concentrations in extremely low gestational age neonates. Pediatr Res. 2022 Jul;92(1):151-167. doi: 10.1038/s41390-021-01814-x. Epub 2021 Nov 30. PMID 34845352
- [Derived] German KR, Vu PT, Comstock BA, Ohls RK, Heagerty PJ, Mayock DE, Georgieff M, Rao R, Juul SE; PENUT Consortium. Enteral Iron Supplementation in Infants Born Extremely Preterm and its Positive Correlation with Neurodevelopment; Post Hoc Analysis of the Preterm Erythropoietin Neuroprotection Trial Randomized Controlled Trial. J Pediatr. 2021 Nov;238:102-109.e8. doi: 10.1016/j.jpeds.2021.07.019. Epub 2021 Jul 27. PMID 34324880
- [Derived] Hingorani S, Schmicker RH, Brophy PD, Heagerty PJ, Juul SE, Goldstein SL, Askenazi D; PENUT Investigators. Severe Acute Kidney Injury and Mortality in Extremely Low Gestational Age Neonates. Clin J Am Soc Nephrol. 2021 Jun;16(6):862-869. doi: 10.2215/CJN.18841220. Epub 2021 Jun 11. PMID 34117080
- [Derived] Mayock DE, Xie Z, Comstock BA, Heagerty PJ, Juul SE; Preterm Epo Neuroprotection (PENUT) Trial Consortium. High-Dose Erythropoietin in Extremely Low Gestational Age Neonates Does Not Alter Risk of Retinopathy of Prematurity. Neonatology. 2020;117(5):650-657. doi: 10.1159/000511262. Epub 2020 Oct 28. PMID 33113526
- [Derived] Juul SE, Vu PT, Comstock BA, Wadhawan R, Mayock DE, Courtney SE, Robinson T, Ahmad KA, Bendel-Stenzel E, Baserga M, LaGamma EF, Downey LC, O'Shea M, Rao R, Fahim N, Lampland A, Frantz ID 3rd, Khan J, Weiss M, Gilmore MM, Ohls R, Srinivasan N, Perez JE, McKay V, Heagerty PJ; Preterm Erythropoietin Neuroprotection Trial Consortium. Effect of High-Dose Erythropoietin on Blood Transfusions in Extremely Low Gestational Age Neonates: Post Hoc Analysis of a Randomized Clinical Trial. JAMA Pediatr. 2020 Oct 1;174(10):933-943. doi: 10.1001/jamapediatrics.2020.2271. PMID 32804205
- [Derived] Askenazi DJ, Heagerty PJ, Schmicker RH, Griffin R, Brophy P, Juul SE, Mayock DE, Goldstein SL, Hingorani S; PENUT Trial Consortium. Prevalence of acute kidney injury (AKI) in extremely low gestational age neonates (ELGAN). Pediatr Nephrol. 2020 Sep;35(9):1737-1748. doi: 10.1007/s00467-020-04563-x. Epub 2020 Jun 2. PMID 32488672
- See also: website for the PENUT Trial — http://PENUT-trial.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Epo 1000 U/kg Followed by 400 U/kg
Started | 464 | 477
Completed | 460 | 476
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Control: Enrollment will occur within 24 hours of birth. Subjects will receive 6 doses of vehicle intravenously during the first 2 weeks of life. Doses will be administered at 48 hour intervals from the time of enrollment. Following high dose administration, sham subcutaneous injections will be given three times a week through to 32-6/7 weeks postmenstrual age. Subjects are then followed until 22-26 months for neurodevelopmental testing.
- Epo 1000 U/kg Followed by 400 U/kg: Enrollment will occur within 24 hours of birth. Epo 1000 U/kg/dose will be administered intravenously for the first 6 doses. Subjects in the Epo arm will then receive 400 U/kg/dose three times a week until they reach 32-6/7 weeks postmenstrual age. Subjects are then followed until 22-26 months for neurodevelopmental testing.
- Total: Total of all reporting groups
Arm/Group | Control | Epo 1000 U/kg Followed by 400 U/kg | Total
Number analyzed (Participants) | 460 | 476 | 936
Age, Customized [Count of Participants; unit: Participants] — Population: Gestational age at birth
  Participants
    24 weeks of gestation | 119 | 113 | 232
    25 weeks of gestation | 124 | 121 | 245
    26 weeks of gestation | 118 | 103 | 221
    27 weeks of gestation | 99 | 139 | 238
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218 | 232 | 450
  Male | 242 | 244 | 486
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 85 | 115 | 200
  Not Hispanic or Latino | 370 | 354 | 724
  Unknown or Not Reported | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 9 | 16
  Asian | 18 | 10 | 28
  Native Hawaiian or Other Pacific Islander | 6 | 2 | 8
  Black or African American | 120 | 120 | 240
  White | 293 | 317 | 610
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 14 | 16 | 30
Region of Enrollment [Number; unit: participants]
  United States | 460 | 476 | 936
Consented and received first study drug dose [Count of Participants; unit: Participants] — Consented subjects who were enrolled according to IRB procedures and who received 1st study drug dose.
  Participants | 460 | 476 | 936

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Death or Severe Neurodevelopmental Impairment (NDI) at 22-26 Months Corrected Age
Description: Severe NDI was defined as Bayley Scales of infant Development, 3rd edition composite motor score or composite cognitive score <70. This instrument is normed at 100 with standard deviation of 15.
  Cerebral palsy was classified as hemiplegia, diplegia, or quadriplegia, and severity was determined according to the Gross Motor Function Classification System (GMFCS) (levels range from 0 [no impairment] to 5 [most severe impairment]). Severe cerebral palsy was defined as a GMFCS level higher than 2.
Time Frame: 22-26 months corrected age
Population: 936 subjects 24-0/7 to 27-6/7 weeks' gestation were randomized and received Epo (n=476) or placebo (n=460) in a double-blinded manner. Survivors who were fully evaluated at 2 years of age are included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Control: Subjects received 6 doses of vehicle intravenously during the first 2 weeks of life. Doses were administered at 48 hour intervals from the time of enrollment. Following high dose administration, sham subcutaneous injections were given three times a week through to 32-6/7 weeks postmenstrual age.
- Epo 1000 U/kg Followed by 400 U/kg: Subjects received 6 doses of intravenous Epo 1000 U/kg/dose at 48 hour intervals from the time of enrollment. Following the high dose period, subjects received subcutaneous Epo 400 U/kg/dose three times a week until 32-6/7 weeks postmenstrual age.
Arm/Group | Control | Epo 1000 U/kg Followed by 400 U/kg
Number analyzed (Participants) | 365 | 376
Participants | 94 | 97
Statistical Analysis 1: Comparison: Control vs Epo 1000 U/kg Followed by 400 U/kg; We evaluated the primary outcome of death or neurodevelopmental impairment using generalized estimating equations to account for potential correlation within siblings from the same pregnancy, with adjustment for gestational age at birth and recruitment site as a fixed effect. The primary analysis included infants with complete data and excluded data from infants known to be alive but in whom neurodevelopmental outcomes were not assessed; Test type: Superiority — We assumed no effect of treatment on death, but that Epo will lead to a decrease in the rate of NDI. If we assume a multiplicative reduction in the NDI rate of 0.45 then we expect a treated NDI rate of 12 percent and an overall rate of death+NDI of 30.4% as compared to the control rate of 40.4% corresponding to an overall treatment rate ratio of 0.75. This leads to a sample size of 376 evaluated subjects per arm or a total evaluated sample size of 752 subjects; p = 0.05, GEE Wald test based on logistic regressi — A two-sided type I error of 0.05 with no formal adjustment for multiple comparisons unless otherwise specified (such as with safety outcomes); adjustments were made for gestational age at birth and recruitment site as a fixed effect; Risk Ratio (RR) = 1.03, .05% CI 2-sided [0.81 to 1.32] — The numerator is the Epo group, denominator is the control group

2. Secondary Outcome: Number of Participants With a Serious Adverse Events (SAE)
Description: Serious adverse events were prespecified. These included any symptomatic thrombosis involving a major vessel, unrelated to an infusion catheter requiring anticoagulation therapy, hematocrit level >65% or an increase of ≥15% in hematocrit in the absence of a preceding blood transfusion, hypertension (defined by receipt of antihypertensive therapy for more than 1 month, discharge with medication, or both), severe pulmonary hemorrhage, severe necrotizing enterocolitis (defined as Bell's stage 2b or 3), severe retinopathy of prematurity resulting in laser surgery or bevacizumab therapy, severe sepsis (defined as culture-proven bacterial or fungal sepsis resulting in blood-pressure support or substantive new respiratory support), grade 3 or 4 intracranial hemorrhage, cardiac arrest that did not result in death, and death.
Time Frame: From birth to hospital discharge (average 12-16 weeks depending on gestational age at birth)
Population: All subjects who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Control: Subjects received 6 doses of vehicle intravenously during the first 2 weeks of life. Doses were administered at 48 hour intervals from the time of enrollment. Following high dose administration, sham subcutaneous injections were given three times a week through to 32-6/7 weeks postmenstrual age (PMA)
- Epo 1000 U/kg Followed by 400 U/kg: Subjects received 6 doses of intravenous Epo 1000 U/kg/dose at 48 hour intervals from the time of enrollment. Following the high dose period, subjects received subcutaneous Epo 400 U/kg/dose three times a week until 32-6/7 weeks postmenstrual age (PMA).
Arm/Group | Control | Epo 1000 U/kg Followed by 400 U/kg
Number analyzed (Participants) | 460 | 476
Participants | 284 | 282
Statistical Analysis 1: Comparison: Control vs Epo 1000 U/kg Followed by 400 U/kg; We hypothesized that Epo would be safe, with no excess of SAEs compared to control infants. Sample size was based on the primary outcome, severe neurodevelopmental impairment or death; Test type: Other — SAEs were defined prospectively. The rate of total SAEs observed through hospital discharge were compared after accounting for potential within-sibship correlation (with multiple gestations) using Generalized Estimating Equations (GEE) with robust standard errors. We used a GEE Wald test based on Poisson or logistic regression for total SAE count and individual events respectively. All other non-categorical data were assessed with GEE regression models appropriate for continuous outcomes; p = 0.05, Poisson regression — Statistical significance was set at 0.05 for the efficacy analysis and for the final safety analysis comparing the rate of total SAEs between treatment groups, and 0.031 for death and 0.004 for the ten individual SAEs due to sequential monitoring; Adjusted for multiple gestation and gestational age; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.83 to 1.22] — Epo is numerator and Control is denominator

3. Secondary Outcome: Imaging
Description: Brain MRI at 36 weeks PMA. Injury scoring was done using a modified scoring system of Kidokoro, with higher scores indicating greater brain injury. Scoring Range: 0-39
Time Frame: 36 weeks postmenstrual age
Population: Patients who survived to 36 weeks postmenstrual age at 9 preselected sites
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Epo 1000 U/kg Followed by 400 U/kg
Number analyzed (Participants) | 101 | 93
score on a scale | 4.1 (2.6) | 3.8 (2.1)
Statistical Analysis 1: Comparison: Control vs Epo 1000 U/kg Followed by 400 U/kg; For all statistical comparisons between groups, Generalized Estimating Equations (GEE) with robust standard errors and a working independence correlation structure for infants included from a multiple gestation were used. A GEE-based Wald test was used to examine differences in the global brain injury severity score between treatment groups, with adjustment for gestational age (GA) at birth used to stratify treatment randomization (24+0 to 25+6 vs. 26+0 to 27+6 in weeks+days of GA); Test type: Superiority; p = 0.36, Generalized estimating equation — Statistical significance was evaluated using a Wald's test and declared significant if p < 0.05; Adjusted for gestational age at birth and treatment assignment

4. Secondary Outcome: Biomarkers
Description: Plasma Epo concentrations were measured in both groups within the first 24 h after birth before study drug administration (baseline), 30 minutes after study drug administration on day 7 (peak Epo concentration) and 30 minutes before study drug on day 9 (trough Epo) and a random level on day 14 after transition to subcutaneous dosing.
Time Frame: Baseline (first 24 hours after birth), days 7, 9 and 14 after birth
Population: Patients who had a baseline Epo level drawn
Measure: Median (Inter-Quartile Range); unit: mU/mL
Groups:
- Control: Subjects received 6 doses of vehicle intravenously during the first 2 weeks of life. Doses will be administered at 48 hour intervals from the time of enrollment. Following high dose administration, sham subcutaneous injections were given three times a week through to 32-6/7 weeks postmenstrual age. Bayley scores of infant development were assessed at 22-26 months
- Epo 1000 U/kg Followed by 400 U/kg: Enrollment occured within 24 hours of birth. Epo 1000 U/kg/dose was administered intravenously for the first 6 doses. Subjects then received 400 U/kg/dose three times a week until 32-6/7 weeks postmenstrual age. Bayley scores of infant development were assessed at 22-26 months
Arm/Group | Control | Epo 1000 U/kg Followed by 400 U/kg
Number analyzed (Participants) | 384 | 391
mU/mL
  Baseline | 7.6 [3.4 to 20.5] | 7 [3.9 to 21.4]
  Peak Epo | 2.2 [1.1 to 4.8] | 2,907 [1,731 to 6998]
  Trough Epo | 5.1 [1.7 to 8.9] | 15.3 [7.4 to 28.9]
  Random (day 14) | 4.6 [2.1 to 8.6] | 25 [9.6 to 66.5]
Statistical Analysis 1: Comparison: Control vs Epo 1000 U/kg Followed by 400 U/kg; For statistical inference, we utilized generalized estimating equations (GEE) with robust standard errors to appropriately account for potential correlation of biomarkers for same-birth siblings. Each respective GEE model adjusted for gestational age at birth and treatment assignment as fixed factors associated with the original study design. Biomarker levels at each follow-up time point were analysed using separate GEE models. Epo levels were log-transformed in all statistical analyses; Test type: Superiority; p < 0.001, Generalized estimating equation — Statistical significance was evaluated using a Wald's test and declared significant if p < 0.007; Adjusted for gestational age at birth and treatment assignment

ADVERSE EVENTS:
Time Frame: Birth to hospital discharge (generally 12 to 16 weeks, depending on gestational age at birth)
Arm/Group | Control | Epo 1000 U/kg Followed by 400 U/kg
All-Cause Mortality (participants affected / at risk) | 45/460 | 53/476
Serious Adverse Events (participants affected / at risk) | 284/460 | 282/476
Other Adverse Events (participants affected / at risk) | 460/460 | 476/476
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=460) | Epo 1000 U/kg Followed by 400 U/kg (N=476)
Polycythemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) — Hematocrit > 65
Major Thrombosis (Blood and lymphatic system disorders) | 2 (2) | 5 (5)
Severe pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 30 (30)
Necrotizing enterocolitis (Gastrointestinal disorders) | 36 (36) | 28 (28)
Severe sepsis (Infections and infestations) | 38 (38) | 35 (35) — Culture positive and symptomatic
Severe intracranial hemorrhage (Nervous system disorders) | 64 (64) | 57 (57) — Grade III or IV
Severe retinopathy of prematurity (Eye disorders) | 30 (30) | 30 (30) — Requiring treatment
Hypertension (Cardiac disorders) | 10 (10) | 6 (6) — Requiring treatment
Nonfatal cardiac arrest (General disorders) | 8 (8) | 9 (9)
Other unexpected life-threatening events (General disorders) | 31 (31) | 27 (27)
Death (General disorders) | 45 (45) | 53 (53)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=460) | Epo 1000 U/kg Followed by 400 U/kg (N=476)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 161 (161) | 172 (172)
Treated patent ductus arteriosus (Cardiac disorders) | 172 (172) | 178 (178)
Necrotizing enterocolitis (Gastrointestinal disorders) | 53 (53) | 46 (46)
Intracranial hemorrhage (all grades) (Nervous system disorders) | 181 (181) | 168 (168)
Periventricular leukomalasia (Nervous system disorders) | 43 (43) | 41 (41)
Cerebellar hemorrhage (Nervous system disorders) | 10 (10) | 8 (8)
Retinopathy of Prematurity (all grades) (Eye disorders) | 258 (258) | 244 (244)
Blood transfusion (Blood and lymphatic system disorders) | 401 (401) | 341 (341)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT01378273/Prot_SAP_000.pdf